CLINICAL TRIAL: NCT00771940
Title: Peripheral Metabolic Effects of Intra Arterial Ghrelin Infusion in Healthy Controls
Brief Title: Peripheral Metabolic Effects of Ghrelin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Jens Otto Lunde Jorgensen/MD Professor and Esben T. Vestergaard/MD PhD, Aarhus University Hospital
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: M-2007008
Record Dates: First submitted 2008-10-08; First posted 2008-10-15 (Estimated); Last update posted 2009-02-03 (Estimated); Status verified 2009-02

CONDITIONS: Healthy Controls
MeSH Terms: interventions — Ghrelin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ghrelin (Active Comparator)
  Interventions: Drug: Ghrelin

INTERVENTIONS:
Drug: Ghrelin — Solvent, cont. infusion

SUMMARY:
The aim of this study is to investigate putative peripheral effects of ghrelin on glucose and lipid metabolism in healthy men. Eight subjects will be enrolled. The hypothesis is that ghrelin infusion causes insulin resistance and lipolysis.

ELIGIBILITY:
Inclusion Criteria:

1. BMI < 27 kg/m2
2. Written informed consent
3. Non-smoker

Exclusion Criteria:

1. Any disease including epilepsy
2. Any use of medications (excl. paracetamol)
3. Present or previous malignancy
4. Alcohol dependency
5. Allergy to any trial medication

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Plasma levels of glucose | During study day

SECONDARY OUTCOMES:
Insulin signaling | Study day
Serum levels of fatty acids | Study day

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L. Jorgensen, MD, Study Director — Medical Department M, Aarhus University Horpital, Denmark; Esben T Vestergaard, PhD, Principal Investigator — Medical Department M, Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark